CLINICAL TRIAL: NCT06558344
Title: A 6-week, Multi-centre, Randomised, Double-blind (Participant and Investigator), Placebo-controlled, Dose-finding Trial to Evaluate the Efficacy, Tolerability, and Safety of Different Doses of Oral BI 1569912 in Patients With Major Depressive Disorder
Brief Title: A Study to Test Different Doses of BI 1569912 in People With Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1447-0012
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BI 1569912 (low dose) (Experimental)
  Interventions: Drug: BI 1569912
- BI 1569912 (medium dose) (Experimental)
  Interventions: Drug: BI 1569912
- BI 1569912 (high dose) (Experimental)
  Interventions: Drug: BI 1569912
- Placebo matching BI 1569912 (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 1569912

INTERVENTIONS:
Drug: BI 1569912 — BI 1569912
  Arms: BI 1569912 (high dose); BI 1569912 (low dose); BI 1569912 (medium dose)
Drug: Placebo matching BI 1569912 — Placebo matching BI 1569912
  Arms: Placebo matching BI 1569912

SUMMARY:
This study is open to adults between 18 and 65 years of age with a type of depression called major depressive disorder. The purpose of the study is to find out whether a medicine called BI 1569912 helps people with depression.

Participants are put into 4 groups randomly, which means by chance. Three of the 4 groups take different doses of BI 1569912 and 1 group takes placebo. Placebo tablets looks like BI 1569912 but do not contain any medicine. Participants take the tablets once a day for 6 weeks.

Participants are in the study for about 2.5 months. During this time, they visit the study site at least 7 times. At the visits, doctors and their staff ask participants about their depression symptoms. At the end of the study, the results are compared between the groups to see whether the treatment works. The doctors also regularly check the general health of participants and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

* Male and female participants, 18 to 65 years of age, both inclusively at the time of consent
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Women of childbearing potential (WOCBP) must be ready and able to use a highly effective method of birth control per ICH M3 (R2) that results in a low failure rate of less than 1% per year when used consistently and correctly plus one additional barrier method. A list of contraception methods meeting these criteria and instructions on the duration of use is provided in the participant information
* Established diagnosis of Major depressive disorder (MDD), single episode or recurrent, as confirmed at the time of screening by the Mini-International Neuropsychiatric Interview (MINI) with a duration of the current depressive episode ≥8 weeks AND ≤24 months at the time of randomisation
* Hamilton Depression Rating Scale-17 (HDRS-17) - Severity scale score ≥20
* Clinical Global Impression- Severity Scale (CGI-S) score ≥4

Exclusion criteria:

* Per Mini International Neuropsychiatric Interview (MINI), have ever met diagnostic criteria for schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar disorder, or delusional disorder
* Diagnosis with antisocial, paranoid, schizoid or schizotypal personality disorder, or MDD with psychotic features as per Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria, at the time of screening visit. Any other personality disorder at screening visit that significantly affects current psychiatric status and likely to impact trial participation, as per the judgement of investigator
* Diagnosis of any other mental disorder that was the primary focus of treatment within 6 months prior to screening (as per clinical discretion of the investigator)
* Treatment failure to 2 or more antidepressants in the current episode, defined as less than 50% response to treatments administered at an adequate dose and duration as evaluated by the Antidepressant treatment response questionnaire (ATRQ)
* History or presence (upon clinical examination) of seizure disorders or an increased risk of seizures (first degree relative with epilepsy), stroke, brain tumour, or any other major neurological illness that could impact participation in the trial
* A current or recent history of clinically significant suicidal ideation with intent within the past 3 months, corresponding to a score of 4 or 5 for ideation on the Columbia-Suicide Severity Rating Scale (C-SSRS) or a suicidal attempt within the past year, as indicated by the C-SSRS at screening visit
* Participants with a body mass index (weight [kg]/height [m]²) lower than 18 kg/m² or greater than 40 kg/m2 at screening
* Diagnosis of a moderate to severe substance related disorder as defined by DSM-5 criteria within 6 months prior to screening visit (with exception of caffeine and tobacco) Further exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in MADRS total score at Week 6 | at baseline and at Week 6
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinician reported interview guide designed to assess the severity of symptoms in depressive illness and to be sensitive to treatment effects.
  The MADRS consists of 10 items:
  1. reported sadness
  2. apparent sadness
  3. inner tension
  4. reduced sleep
  5. reduced appetite
  6. concentration difficulties
  7. lassitude
  8. inability to feel
  9. pessimistic thought
  10. suicidal thoughts
  Symptoms are rated on a 7-point Likert scale from 0 (no symptom) to 6 (severe symptom).
  Definitions of severity are provided at 2-point intervals. The possible total score could range from 0 to 60 (from normal with absence of symptoms to severe depression).

CONTACTS AND LOCATIONS:
Locations (41):
- United States (35):
  - Clinical Innovations, Inc, Bellflower, California
  - ASCLEPES Research Centers, P.C. dba Alliance Research, Long Beach, California
  - Excell Research Inc., Oceanside, California
  - CiTrials-Riverside-63180, Riverside, California
  - Artemis Institute for Clinical Research, LLC, San Diego, California
  - Lumos Clinical Research, San Jose, California
  - California Neuroscience Research, Sherman Oaks, California
  - Pacific Clinical Research Management Group LLC, Upland, California
  - Research Centers of America-Hollywood-67537, Hollywood, Florida
  - Clinical Neuroscience Solutions, Inc-Jacksonville-62642, Jacksonville, Florida
  - CCM Clinical Research Group, LLC-Miami-68482, Miami, Florida
  - Optimus U Corporation-Miami-69452, Miami, Florida
  - Clinical Neuroscience Solutions, Inc-Orlando-62685, Orlando, Florida
  - Advanced Discovery Research LLC, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Psych Atlanta, PC, Marietta, Georgia
  - Pharmasite Research, Incorporated, Baltimore, Maryland
  - Copley Clinical, Boston, Massachusetts
  - Boston Clinical Trials, Roslindale, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - ActivMed, Portsmouth, New Hampshire
  - Center For Emotional Fitness, Cherry Hill, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Integrative Clinical Trials LLC, Brooklyn, New York
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Berman Clinical, New York, New York
  - Davis Clinical, The Bronx, New York
  - Sooner Clinical Research, Inc, Oklahoma City, Oklahoma
  - Surburban Research Associates, Inc., Media, Pennsylvania
  - Clinical Neuroscience Solutions, Inc-Memphis-65988, Memphis, Tennessee
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Core Clinical Research, Everett, Washington
- Japan (6):
  - Uematsu Mental Clinic, Fukuoka, Chikugo
  - Kaku Mental Clinic, Fukuoka, Fukuoka
  - Hirota Clinic, Fukuoka, Kurume
  - Yutaka Clinic, Kanagawa,Sagamihara
  - Maynds Tower Mental Clinic, Tokyo, Shibuya-ku
  - Ichigaya Himorogi Clinic, Tokyo, Shinjuku-ku

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com